CLINICAL TRIAL: NCT04598048
Title: Quality of Life Post-ACS in Participants from EMMACE
Acronym: EMMACE-XL
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Dr Christopher Gale, Professor of Cardiovascular Medicine, University of Leeds
Other Study IDs: 20/PR/0104; 276202 (Other: IRAS); PG/19/54/34511 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2020-10-07; First posted 2020-10-22 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- EMMACE 3: Participants who were recruited to the EMMACE 3 study and have agreed to contact for further research.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Patients will complete an EQ-5D questionnaire, medication and lifestyle questions

SUMMARY:
EMMACE-XL will recruit participants who are survivors of acute coronary syndrome (a type of heart attack) to assess their health-related quality of life five years or more after their heart attack. We will invite surviving participants from the EMMACE 3 and 4 studies to consent to participate in EMMACE-XL study, they will be asked to complete one questionnaire relating to their health, medication and lifestyle. The questionnaire will be linked to their data collected as part of the EMMACE 3 and 4 studies including long term follow up data from NHS Digital.

The data collected from all the studies will then be analysed to see if patient groups can be identified who are at risk of poorer quality of life and worse health outcomes. These groups can then be targeted with the aim of improving their health outcomes.

The study will use statistical methods to look at the relationship of factors such as; medication adherence, comorbidities and patient demographics on health-related quality of life and health outcomes.

DETAILED DESCRIPTION:
Health-related quality of life (HRQoL) after myocardial infarction (MI) is an important clinical outcome. It allows the definition of health outcomes from a patient's perspective and, therefore, offers the potential to collect patient-centered ill-health, which may be used as an additional endpoint in the evaluation of care. Many survivors of MI experience poor HRQoL, and many patients consider the quality of additional life years gained just as important as the length of life. The goal of contemporary therapies, therefore, should be not only to extend life expectancy, but also to ensure a high quality long-term health state. Accordingly, HRQoL is increasingly being used as an outcome measure in clinical trials evaluating both the impact of disease burden and the effectiveness of cardiovascular interventions.

Research has shown that changes in HRQoL are associated with a range of clinical outcomes, including death, anxiety and depression, and medications compliance. Changes in HRQoL have been reported to negatively impact healthcare costs, and employment. However, there is a paucity of information about the relationship between HRQoL and clinical outcomes inherent following MI. Moreover, previous research is limited by small sample sizes, poor generalisability,selection bias, the use of retrospective cross-sectional designs,and short follow-up durations of 6 months - 2 years. For example in our previous studies (EMMACE 3 and 4 ), we followed up patients for up to 2 years. The EMMACE data analysis showed that over two years HRQoL improved for the majority (two thirds) but was significantly worse and more likely to decline for women, NSTEMI, and people with long-term health conditions .

Whilst the analysis of EMMACE demonstrates promising results, the EMMACE data are limited by the short follow up period of up to 2 years. We have been funded by the British Heart Foundation (Program grant number PG/19/54/34511) to link the EMMACE 3 and 4 data to ONS (mortality) and Hospital Episode Statistics (HES) data such that longer-term non-fatal and fatal outcomes and healthcare utilisation may be studied. All patients were consented to enter the EMMACE 3 and 4 studies and for their self-reported data to be linked to future electronic health record data. EMMACE data has already been successfully linked to data from the national heart attack registry (Myocardial Ischemia National Audit project, MINAP) thus providing information about hospital treatment for MI and comorbidities. This study will provide a further follow up of this data so that longer term follow up can be studied.

To complement our work, and given the paucity on longer term HRQoL data, in this proposal we aim to collect > 5 years HRQoL measures data from the participants of EMMACE 3 & 4 studies. The longer follow up of HRQoL data (> 5 years) may provide insights into understanding the association between long term changes in HRQoL and subsequent clinical outcomes and precisely in whom worse (or better) outcomes may occur will permit the design and testing of novel intervention to reduce premature death from MI.

The planned research will provide unique and comprehensive insight into the relationship between changes in HRQoL and survival following MI. Health-related quality of life is a patient reported outcome measure (PROM) which can detect change in risk of events for patients, and potentially serve as a predictor of future risk (using patient-facing data capture tools). Understanding the association between changes in HRQoL and health outcomes and precisely in whom worse (or better) outcomes may occur will permit the design and testing of novel interventions to reduce premature death from MI.

ELIGIBILITY:
Inclusion Criteria:

Surviving participants of the EMMACE 3 & 4 studies, who have agreed to be contacted for further research

Exclusion Criteria:

Concerns by the research team of mental capacity.

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Surviving participants of the EMMACE 3 & 4 studies.
  Participants of the EMMACE 3 and 4 studies were recruited between November 2011 and June 2015 following a heart attack and admission to a UK hospital
Sampling Method: Probability Sample
Enrollment: 13400 (Actual)
Dates: Start 2020-09-27 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
To describe ACS patients according to their changes in HRQoL trajectory and determine factors associated with poor HRQoL. | From first recruited into data received - approx 10 years
  Surviving ACS patients recruited in the EMMACE 3 and 4 studies and have consented to further contact will be contacted and requested to completed a EQ-5D questionnaire. Sequential EQ-5D-3L and EQVAS data will be used both as a measure of outcome (recovery pattern) and predictor of outcome. Multilevel modelling will be used to determine factors associated with poor HRQoL.
  The study will use statistical modelling approaches to investigate the relationship of factors such as; medication adherence, co-morbidities and patient demographics on health-related quality of life and health outcomes. This will help identify patient groups at risk of poorer quality of life and worse outcomes to enable these groups to be targeted to improve their outcomes.

SECONDARY OUTCOMES:
To investigate the association between changes in HRQoL and mortality post ACS. | From first recruited into data received - approx 10 years
  Surviving ACS patients recruited in the EMMACE 3 and 4 studies and have consented to further contact will be contacted and requested to completed a EQ-5D questionnaire. The data will also be linked to mortality data supplied by ONS. Sequential EQ-5D-3L and EQVAS data will be used both as a measure of outcome (recovery pattern) and predictor of outcome. Joint modelling of changes in HRQoL and survival will be used to investigate the association of HRQoL and mortality.
To summarise the incidence of fatal and non-fatal health outcomes amongst our patients and determine if there are common patient clusters with respect to these outcomes. | From first recruited into data received - approx 10 years
  We will use mortality and hospital episodes data for all patients recruited to the EMMACE 3 and 4 studies to compare their fatal and non fatal health outcomes to see if there are any common patient clusters with respect to these outcomes.
To investigate the association of quality of care, cardiac rehabilitation, medications, patient characteristics, socioeconomic status, changes in HRQoL with mortality | From first recruited into data received - approx 10 years
  We will combine mortality, hospital episodes data, EQ-5D and medication adherence responses from surviving ACS patients for the EMMACE 3 and 4 studies who have consent to further follow up to investigate whether there is any associations between quality of care, cardiac rehabilitation, medications, patient characteristics, socioeconomic status, changes in HRQoL with mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Chris P Gale, Prof, Principal Investigator — University of Leeds
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared as per patient consent.

REFERENCES:
- [Background] Alabas OA, West RM, Gillott RG, Khatib R, Hall AS, Gale CP; EMMACE-3 Investigators. Evaluation of the Methods and Management of Acute Coronary Events (EMMACE)-3: protocol for a longitudinal study. BMJ Open. 2015 Jun 23;5(6):e006256. doi: 10.1136/bmjopen-2014-006256. PMID 26105029
- [Background] Munyombwe T, Hall M, Dondo TB, Alabas OA, Gerard O, West RM, Pujades-Rodriguez M, Hall A, Gale CP. Quality of life trajectories in survivors of acute myocardial infarction: a national longitudinal study. Heart. 2020 Jan;106(1):33-39. doi: 10.1136/heartjnl-2019-315510. Epub 2019 Nov 7. PMID 31699696
- [Derived] Dondo TB, Munyombwe T, Hall M, Hurdus B, Soloveva A, Oliver G, Aktaa S, West RM, Hall AS, Gale CP. Sex differences in health-related quality of life trajectories following myocardial infarction: national longitudinal cohort study. BMJ Open. 2022 Nov 8;12(11):e062508. doi: 10.1136/bmjopen-2022-062508. PMID 36351712
- See also: Activities of the team and link to study information — https://lida.leeds.ac.uk/research-projects/566-2/